CLINICAL TRIAL: NCT04146766
Title: Effectiveness of eHealth on the Self-management, Physiological Health and Quality of Life Among Coronary Artery Disease Patients
Brief Title: Effectiveness of eHealth on the Self-management of Health Status and QOL Among CAD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hui-Hsun Chiang, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2-108-05-132
Record Dates: First submitted 2019-10-22; First posted 2019-10-31 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: eHealth; Coronary Artery Disease; Quality of Life; Self-management
Keywords: Coronary artery disease; Remote Care; artificial intelligence; self-management; Quality of Life
MeSH Terms: conditions — Coronary Artery Disease | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: wait list control group RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth (Experimental): Provide home physiology measurement services, including automatic uploading of measured blood pressure values to the cloud, serial back-end education platform to provide numerical anomaly alarms and health care notifications, monthly measurement data reports, combined with mobile APP management system for immediate enquiry . In addition to the electric visit to the patient's health education guidance, the content includes: 1. Encourage the walking exercise to perform 2. Ask the walking exercise execution progress, please return the daily value of the case to facilitate the record 3. Answer the relevant questions asked during the intervention.
  Interventions: Combination Product: eHealth
- wait list control (Experimental): wait list control for 3 months and then Provide home physiology measurement services, including automatic uploading of measured blood pressure values to the cloud, serial back-end education platform to provide numerical anomaly alarms and health care notifications, monthly measurement data reports, combined with mobile APP management system for immediate enquiry . In addition to the electric visit to the patient's health education guidance, the content includes: 1. Encourage the walking exercise to perform 2. Ask the walking exercise execution progress, please return the daily value of the case to facilitate the record 3. Answer the relevant questions asked during the intervention.
  Interventions: Combination Product: eHealth

INTERVENTIONS:
Combination Product: eHealth — The study was randomized (wait-list-control), and it was estimated that 60 subjects were randomly assigned to the immediate treatment group and the wait-list-control group. The two groups were tested for baseline before intervention in the eHealth. After the first questionnaire evaluation, the experimental group was involved in the eHealth for three months, and after three months, the experimental group and the waiting intervention control group were post-tested. To assess the effectiveness of the two groups before and after the eHealth . Control group that waits for intervention in the fourth month from the beginning of the fourth month to the end of the sixth month

SUMMARY:
This article uses the smart medical case management tracking system, combined with various terminal devices to fully record the measured data (pulse, blood pressure) for case home care tracking to prevent the occurrence and deterioration of the disease. Therefore, with the promotion of the eHealth medical staff and members of the family can instantly grasp the health of the body and cultivate the habits of self-health management and enhance the quality of care. Therefore, we hope to use the Smart Health Cloud as an interventional measure to improve the care of patients with coronary artery disease, improve self-management ability and quality of life.

DETAILED DESCRIPTION:
The World Health Organization points out that cardiovascular disease is the number one killer of global deaths, killing 17.1 million people worldwide each year, accounting for 31% of the world's total deaths. Heart disease is the second leading cause of death in China. Coronary artery disease (CAD) is the majority, and coronary artery disease is the most common cardiovascular disease. Good self-management can reduce disease risk factors and improve related prognosis. It is also an important issue in health promotion around the world. This article uses the smart medical case management tracking system, combined with various terminal devices to fully record the measured data (pulse, blood pressure) for case home care tracking to prevent the occurrence and deterioration of the disease. Therefore, with the promotion of the eHealth medical staff and members of the family can instantly grasp the health of the body and cultivate the habits of self-health management and enhance the quality of care. Therefore, we hope to use the Smart Health Cloud as an interventional measure to improve the care of patients with coronary artery disease, improve self-management ability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* A patient who is 20 years of age or older and has a Coronary computed tomography angiography >50% vascular stenosis, has been PTCA、stent or CABG
* Taiwanese, understand Chinese

Exclusion Criteria:

* Those who can't express their wishes clearly (such as Azheimer's disease, mental dysfunction)
* mental disorder
* infectious diseases
* Patients who participate in other research projects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
physiological indicators-HDL-C(T1) | T1-baseline
  HDL-C, the unit is mg/dL
physiological indicators-HDL-C(T2) | T2-three months later
  HDL-C, the unit is mg/dL
physiological indicators-HDL-C(T3) | T3-six months later
  HDL-C, the unit is mg/dL
physiological indicators-LDL-C(T1) | T1-baseline
  LDL-C, the unit is mg/dL
physiological indicators-LDL-C(T2) | T2-three months later
  LDL-C, the unit is mg/dL
physiological indicators-LDL-C(T3) | T3-six months later
  LDL-C, the unit is mg/dL
physiological indicators-Total Cholesterol(T1) | T1-baseline
  Total Cholesterol, the unit is mg/dL
physiological indicators-Total Cholesterol(T2) | T2-three months later
  Total Cholesterol, the unit is mg/dL
physiological indicators-Total Cholesterol(T3) | T3-six months later
  Total Cholesterol, the unit is mg/dL
physiological indicators-Triglyceride(T1) | T1-baseline
  Triglyceride, the unit is mg/dL
physiological indicators-Triglyceride(T2) | T2-three months later
  Triglyceride, the unit is mg/dL
physiological indicators-Triglyceride(T3) | T3-six months later
  Triglyceride, the unit is mg/dL
physiological indicators-GLU(T1) | T1-baseline
  GLU, the unit is mg/dL
physiological indicators-GLU(T2) | T2-three months later
  GLU, the unit is mg/dL
physiological indicators-GLU(T3) | T3-six months later
  GLU, the unit is mg/dL
physiological indicators-HbA1C(T1) | T1-baseline
  HbA1C, the unit is %
physiological indicators-HbA1C(T2) | T2-three months later
  HbA1C, the unit is %
physiological indicators-HbA1C(T3) | T3-six months later
  HbA1C, the unit is %

SECONDARY OUTCOMES:
self-management-T1 | T1-baseline
  use The partners in Health scale. total of 12 questions,The scoring method uses the nine-point Likert Scales score. The score of 0 is divided into self-management performance, and the score of 8 indicates that self-management is good. The total score is 96 points. The higher the score, the better the self-management.
self-management-T2 | T2-three months later
  use The partners in Health scale. total of 12 questions,The scoring method uses the nine-point Likert Scales score. The score of 0 is divided into self-management performance, and the score of 8 indicates that self-management is good. The total score is 96 points. The higher the score, the better the self-management.
self-management-T3 | T3-six months later
  use The partners in Health scale. total of 12 questions,The scoring method uses the nine-point Likert Scales score. The score of 0 is divided into self-management performance, and the score of 8 indicates that self-management is good. The total score is 96 points. The higher the score, the better the self-management.

OTHER OUTCOMES:
Quality of life scale-T1 | T1-baseline
  use WHOQOL-BREF Taiwan Version. total of 28 questions,The scoring method uses the five-point Likert Scales score The questionnaire has a total of 28 questions, with at least one point for each question and a maximum of five points. The higher the score, the better the quality of life.
Quality of life scale-T2 | T2-three months later
  use WHOQOL-BREF Taiwan Version. total of 28 questions,The scoring method uses the five-point Likert Scales score The questionnaire has a total of 28 questions, with at least one point for each question and a maximum of five points. The higher the score, the better the quality of life.
Quality of life scale-T3 | T3-six months later
  use WHOQOL-BREF Taiwan Version. total of 28 questions,The scoring method uses the five-point Likert Scales score The questionnaire has a total of 28 questions, with at least one point for each question and a maximum of five points. The higher the score, the better the quality of life.
Modified Health care machine rating scale | T2-three months later
  There are three questions in the satisfaction survey. Use category options to measure usage satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- TSGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No